CLINICAL TRIAL: NCT00476008
Title: Delaying the Progression of Driving Impairment in Individuals With Mild Alzheimer's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Florida Atlantic University (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NAM-MD-49
Record Dates: First submitted 2007-05-17; First posted 2007-05-21 (Estimated); Results first posted 2014-06-03 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-08

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; Mild Alzheimer's Disease; Driving; Driving Impairment
MeSH Terms: conditions — Alzheimer Disease | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): One tablet placebo morning and evening (BID) for 12 months
  Interventions: Drug: Placebo
- Memantine (Active Comparator): One tablet memantine (Namenda)10mg morning and evening (BID) for 12 months.
  Interventions: Drug: Memantine

INTERVENTIONS:
Drug: Memantine — One tablet memantine (Namenda)10mg morning and evening (BID) for 12 months
  Other Names: Namenda
  Arms: Memantine
Drug: Placebo — One tablet placebo morning and evening (BID) for 12 months
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine whether memantine delays the progression of driving impairment in patients with mild Alzheimer's Disease (AD).

DETAILED DESCRIPTION:
It is well known, and of great concern to both patients and families, that individuals with Alzheimer's disease (AD) eventually become driving impaired. Drivers with dementia are estimated to be 2-8 times more likely to be involved in an automobile crash as unimpaired peers. Approximately half of individuals with mild AD have the skills needed to drive safely. Formal driver evaluation may be necessary to make this distinction. Some reviews in the literature have suggested that individuals identified as high risk, such as those with AD, be advised by their physicians to cease driving altogether. Other studies suggest that these individuals may continue to drive for up to 4 years following diagnosis. Memantine may be effective in delaying the progression of driving impairment in individuals with mild AD. If the investigators can demonstrate a significant delay in the decline in the driving ability, this could extend their driving time and therefore be of immense benefit to patients and their caregivers.

Comparison(s): Subjects treated with memantine over a period of 12 months, compared to subjects on placebo.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 60 years of age and older
* Subjects must either be previously diagnosed with mild Alzheimer's Disease (AD) by a neurologist, psychiatrist, geriatrician, or be evaluated at a Memory Disorders Center prior to entry into the study
* Subjects must have a score of ≥ 23 on the Mini-Mental State Examination (MMSE) at the Screening Visit
* Subjects must receive a passing score on the DriveABLE test
* Female subjects must be at least 2 years post-menopausal or surgically sterile
* Written informed consent must be obtained from the subject prior to the initiation of any study specific procedures

Exclusion Criteria:

* Subjects who have been treated with a depot neuroleptic within six (6) months of the Screening Visit
* Subjects who fail the OPTEC vision test at the screening visit
* Subjects who score > 7 on the Hachinski Test at the screening visit
* Subjects with evidence of clinically significant and active pulmonary, gastrointestinal, renal, hepatic, endocrine or cardiovascular system disease (subjects with controlled hypertension, right bundle branch block [complete or partial] and pacemakers may be included in the study). Subjects with thyroid disease may also be included in the study, provided they are euthyroid on treatment. Subjects with controlled diabetes may also be included
* Recent (< 2years) B12 or folate deficiency that was considered clinically significant
* Subjects with evidence of other psychiatric/neurologic disorders including, but not limited to, stroke, Vascular Dementia, Lewy-Body Disease, Parkinson's Disease, seizure disorder, head injury with loss of consciousness within the past 5 years, any psychotic disorder, or bipolar disorder
* Subjects who are taking, or have taken, amantadine, ketamine, dextromethorphan that cannot be discontinued or switched to an allowable alternative medication prior to the minimum allowable interval before Baseline
* Subjects who have been in an investigational drug study or who have received treatment with an investigational drug within 30 days (or 5 half-lives, whichever is longer) of the Screening Visit
* Any condition, which would make the subject, in the opinion of the investigator, unsuitable for the study
* If subjects are taking Acetylcholinesterase inhibitors (AChEls), they must be on a stable dose for > 3 months prior to baseline. No initiation of AChEls is permitted; discontinuation and dose reduction are permitted

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-07; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Holland, MD, Principal Investigator — Charles E, Schmidt College of Medicine at Florida Atlantic University
Locations (1):
- Charles E. Schmidt College of Medicine, Florida Atlantic University, Boca Raton, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment dates July 2007 - September 2011 Newspaper print ads, physician referral, subject referral, press releases
Pre-assignment Details: Prior to randomization, subjects completed a screening visit to discuss/sign informed consent and determine study eligibility. Of the 60 subjects screened, 17 were excluded due to not passing the screening visit driving test, scoring out of the inclusion criteria range on screening visit assessments or meeting an exclusion criteria.
Groups:
- Memantine: Memantine : Memantine (Namenda)10mg BID for 12 months
- Placebo: Placebo : Placebo BID for 12 months
Period: Overall Study
Arm/Group | Memantine | Placebo
Started | 22 | 21
6 Month Testing | 15 | 14
Completed | 13 | 13
Not Completed | 9 | 8
Not completed — Adverse Event | 4 | 4
Not completed — Placebo concerns | 2 | 2
Not completed — Physician Decision: Medication Noncompli | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Memantine | Placebo | Total
Number analyzed (Participants) | 22 | 21 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 21 | 21 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.13 (6.38) | 80.47 (5.92) | 79.28 (6.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 15
  Male | 12 | 16 | 28
Region of Enrollment [Number; unit: participants]
  United States | 22 | 21 | 43

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Measure is the Number of Subjects in Each Group Who Are Able to Pass the DriveABLE On-Road Test at Month 12 (Endpoint).
Description: The DriveABLE On-Road Test utilizes a standardized road course and standardized scoring procedures designed to identify driving errors indicative of decline in competence scores. This road test takes approximately 30-45 minutes and covers a distance of approximately 9 miles.
Time Frame: Baseline and 12 months
Population: One subject in the placebo group could not complete the driving test at 12 months due to his vision being below the legal limit to drive.
Measure: Number; unit: participants
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 13 | 12
participants
  DriveABLE passed | 13 (0) | 10
  DriveABLE same or improved | 13 | 9

2. Secondary Outcome: Fuld Object Memory Evaluation
Description: Ten common objects in a bag were presented to determine whether the subject could identify objects by touch. The subject was not told that memory of this event would be tested. The subject names each object and then pulls it out of the bag to see if he is correct. After distracting the subject, by asking the patient to say words rapidly from a single category (rapid verbal retrieval), the subject is asked to recall the objects from the bag. The subject was then offered two more chances to learn and recall them (store and retrieve) by reminding the subject of omitted items after each recall, with rapid verbal retrieval preventing rehearsal before each recall opportunity.
  Retrieval scores were summed over the three trials with the range of possible scores being 0-30. Lower scores indicate more severe impairment.
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 13 | 13
units on a scale
  Baseline Sum of Retrieval Score | 18.87 (5.00) | 18.38 (8.76)
  12 month Sum of Retrieval Score | 19.08 (8.47) | 17.94 (5.85)

3. Secondary Outcome: Rey Complex Figure Test
Description: This is a measure of visual-spatial and constructional ability as well as higher order cognitive processes including planning, organizing, and problem solving. Subjects are asked to copy a complicated drawing. 18 elements are scored from 0-2 depending on accuracy/distortion and location of the reproduction. The maximum score is 36 points. Lower scores indicate more severe impairment
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 13 | 13
units on a scale
  Baseline | 27.53 (6.05) | 29.30 (5.10)
  12 Months | 29.96 (4.54) | 27.85 (5.75)

4. Secondary Outcome: Trail Making Test - Part A
Description: A simple test of visual tracking. The score is the time in seconds required to complete. Higher scores indicate lower functioning.
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 13 | 13
seconds
  Baseline | 50.33 (17.2) | 39.63 (12.37)
  12 months | 53.46 (22.00) | 38.54 (16.32)

5. Secondary Outcome: Trail Making Test - Part B
Description: This tests cognitive flexibility and set-shifting. It is considered to be a test of executive functioning and has been shown to correlate with on-road driving ability. The score is the time in seconds required to complete each part. Higher scores indicate decreased functioning.
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 13 | 13
seconds
  Baseline | 195.33 (128.58) | 117.75 (43.03)
  12 months | 233.15 (159.49) | 170.92 (145.33)

6. Secondary Outcome: Mini Mental Status Exam
Description: Scores range from 0-30 with lower scores indicating decreased functioning.
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 13 | 13
units on a scale
  Baseline | 27.67 (1.63) | 28.13 (2.00)
  12 Months | 26.00 (3.56) | 27.15 (2.34)

7. Secondary Outcome: Useful Field of View
Description: The Useful Field of View is a computer-administered test that measures higher order processing skills such as divided attention and visual processing speed. Scores can be predictive of ability to perform many everyday activities, such as driving a vehicle. Speed of visual processing is measured as the examinee identifies a target, but must also localize a simultaneously presented target displayed in the periphery of the computer monitor. Scores range from 1 to 4 with 1 being no impairment, 2= mild, 3= moderate and 4=serious impairment.
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 13 | 13
units on a scale
  Baseline | 3.00 (1.31) | 2.44 (1.50)
  12 months | 2.54 (1.45) | 2.08 (1.38)

8. Secondary Outcome: Motor Free Visual Perception Test - Visual Closure Subtest
Description: This is an 11 item multiple choice test of visual perception. Scores range from 0-11. This test measures visual perception deficits separate from motor skill abilities. Higher scores indicate more severe impairment.
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: number incorrect
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 13 | 13
number incorrect
  Baseline | 2.93 (2.52) | 2.00 (2.19)
  12 months | 3.23 (2.83) | 2.69 (2.53)

9. Secondary Outcome: Cognitive Dementia Rating Scale
Description: This scale is used to stage severity of dementia. Scores are on a five-point scale in which 0 indicates no cognitive impairment, .5 = very mild dementia,1 = mild, 2 = moderate and 3= severe.
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 13 | 13
units on a scale
  Baseline | 2.30 (1.31) | 2.41 (1.11)
  12 Months | 2.31 (2.71) | 1.81 (1.61)

10. Secondary Outcome: Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog)
Description: The ADAS-Cog is a performance based test that measures specific cognitive and behavioral dysfunctions in patients with Alzheimer's disease. The cognitive subscale comprises 11 items which measure word recall (0-10), ability to follow single and multi-step commands (0-5), constructional praxis (0-5), ideational praxis (0-5), naming objects(0-5), word recognition (0-12), orientation (0-8), comprehension of spoken language (0-5), word finding difficulty(0-5) and ability to remember test instructions (0-5). 0 = no impairment with higher scores indicating more severe impairment.
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 13 | 13
units on a scale
  1) Word Recall - Baseline | 4.33 (1.28) | 4.00 (1.26)
  1) Word Recall - 12 Months | 4.56 (1.97) | 4.13 (1.31)
  2) Commands - Baseline | .40 (.51) | 0 (0)
  2) Commands - 12 Months | .23 (.60) | .85 (2.76)
  3) Constructional Praxis - Baseline | 3.40 (.51) | 3.44 (.63)
  3) Constructional Praxis - 12 Months | 3.54 (.52) | 3.46 (.52)
  4) Ideational Praxis - Baseline | 5.00 (0) | 5.00 (0)
  4) Ideational Praxis - 12 months | 4.92 (.28) | 5.00 (0)
  5) Naming - Baseline | 1.80 (1.70) | 2.38 (3.93)
  5) Naming - 12 months | 1.31 (1.38) | 1.77 (1.69)
  6) Orientation - Baseline | .80 (1.01) | .44 (1.09)
  6) Orientation - 12 Months | .85 (1.34) | .46 (.88)
  7) Word Recognition - Baseline | 9.60 (6.07) | 7.27 (5.42)
  7) Word Recognition - 12 Months | 8.10 (8.39) | 9.31 (4.91)
  8) Remember Test Instructions - Baseline | 0.00 (0) | 0.00 (0)
  8) Remember Test Instructions - 12 Months | 0.00 (0) | 0.00 (0)
  9) Spoken Language - Baseline | .20 (.77) | 0.00 (0)
  9) Spoken Language - 12 Months | .23 (.83) | 0 (1.00)
  10) Word Finding - Baseline | .13 (.52) | 0.00 (0)
  10) Word Finding - 12 Months | .15 (.55) | .08 (.28)
  11) Comprehension - Baseline | .07 (.26) | .06 (.25)
  11) Comprehension - 12 Months | .31 (.63) | .15 (.38)

ADVERSE EVENTS:
Arm/Group | Memantine | Placebo
Serious Adverse Events (participants affected / at risk) | 2/22 | 3/21
Other Adverse Events (participants affected / at risk) | 6/22 | 9/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Memantine (N=22) | Placebo (N=21)
Mouth Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Generalized Weakness (General disorders) | 0 (0) | 1 (1)
Stroke (Vascular disorders) | 0 (0) | 1 (1)
Rectal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Memantine (N=22) | Placebo (N=21)
Dizziness (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 4 (4) | 3 (3)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Decreased Appetite (Gastrointestinal disorders) | 2 (2) | 0 (0)
Insomnia (Nervous system disorders) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (3)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes